CLINICAL TRIAL: NCT06166823
Title: Electronic Medical Record Alerts to Optimize Medical Therapy in Heart Failure and Reduced Ejection Fraction in a Low-middle Income Country
Brief Title: Electronic Medical Record Alerts to Optimize Medical Therapy in Heart Failure and Reduced Ejection Fraction
Acronym: OPTIMAL-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Cardiovascular de Buenos Aires (Other)
Responsible Party: Principal Investigator, Lucrecia Maria Burgos, MD, Instituto Cardiovascular de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: HFrEF - Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMR Alert (Experimental)
  Interventions: Other: EMR alert
- Usual Care (No Intervention)

INTERVENTIONS:
Other: EMR alert — EMR alert for medication optimization
  Arms: EMR Alert

SUMMARY:
OPTIMAL-HF is a pragmatic, cluster randomized, single-blind intervention trial that will be conducted at an outpatient clinic in Argentina. The trial will assess the effectiveness of an individualized-based alert system compared to usual care in improving GDMT optimization at 90 days in patients with HFrEF.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Eligible patients will include those with an EF ≤ 40% on their most recent echocardiogram, age > 18, and an outpatient cardiology encounter during the study period.
* Age 18 or over

Exclusion Criteria:

* under optimal medical treatment
* palliative care, or undergoing hemodialysis will be excluded

Cardiologist

Inclusion criteria:

Cardiologists from an outpatient clinic at a cardiovascular center in Buenos Aires will be selected for potential participation in the study.

Exclusion criteria Cardiologists belonging to the heart failure service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the GDMT optimize score in HfrEF patients 90 days after randomization. | 90 days

IPD SHARING:
Plan to Share IPD: Undecided